CLINICAL TRIAL: NCT06542198
Title: Mannitol-induced Release of Copeptin in Healthy Adults and Patients With Polyuria-Polydipsia Syndrome: a Double-blind, Randomized Crossover Proof-of-concept and Open-label Single Arm Pilot Study (MARS Study)
Brief Title: Mannitol-induced Release of Copeptin in Healthy Adults and Patients With Polyuria-Polydipsia Syndrome (MARS Study)
Acronym: MARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-01214; kt24ChristCrain
Record Dates: First submitted 2024-07-26; First posted 2024-08-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Polyuria-polydipsia Syndrome; Arginine Vasopressin Deficiency; Primary Polydipsia
Keywords: Hypertonic saline infusion; Mannitol; Copeptin
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Polydipsia, Psychogenic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: The study is conducted in two parts. Part 1: Cross-over proof-of-concept study Part 2: Single arm case-control pilot study
Masking Description: The study is conducted in two parts. Part 1: Double-blind Part 2: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy adults (Experimental): Part 1 of the study is conducted with healthy adults.
  Interventions: Diagnostic Test: Mannitol Infusion (blinded); Diagnostic Test: Placebo Infusion (blinded)
- Primary polydipsia (PP) patients (Experimental): Part 2 of the study is conducted with PP patients.
  Interventions: Diagnostic Test: Mannitol Infusion (open label)
- Arginine vasopressin deficiency (AVP-D) patients (Experimental): Part 2 of the study is conducted with AVP-D patients.
  Interventions: Diagnostic Test: Mannitol Infusion (open label)

INTERVENTIONS:
Diagnostic Test: Mannitol Infusion (blinded) — 1 g of mannitol per kg body weight is infused in 30 minutes (≙ 5 ml/kg body weight), with an upper limit of 80 g, equivalent to a body weight of 80 kg or a volume of 400 ml. The solution used for infusion is 20% mannitol in water for injection and is administered at a rate of 0.17 ml/kg/min.
  Arms: Healthy adults
Diagnostic Test: Placebo Infusion (blinded) — 0.9% saline will be administered in the same amount as the mannitol dose infusion (= 5 ml/kg body weight), with a rate of 0.17 ml/kg/min in 30 minutes, with an upper limit of 400 ml (equivalent to a body weight of 80 kg).
  Arms: Healthy adults
Diagnostic Test: Mannitol Infusion (open label) — 1.5 g of mannitol per kg body weight is infused in 30 minutes (≙ 7.5 ml/kg body weight), with an upper limit of 120 g, equivalent to a body weight of 80 kg or a volume of 600 ml. The solution used for infusion is 20% mannitol in water for injection.
  Arms: Arginine vasopressin deficiency (AVP-D) patients; Primary polydipsia (PP) patients

SUMMARY:
The aims of this study are to investigate whether mannitol stimulates copeptin (part 1: proof-of-concept) and whether the copeptin levels upon mannitol infusion differ in primary polydipsia and arginine vasopressin deficiency (part 2: pilot study).

DETAILED DESCRIPTION:
Diagnosing polyuria-polydipsia syndrome, which includes arginine vasopressin (AVP) deficiency (AVP-D, formerly central diabetes insipidus) and primary polydipsia (PP), is challenging but essential. Currently, the most accurate test currently involves measuring copeptin after osmotic stimulation with hypertonic saline, but this test is rarely used due to the need for close sodium monitoring and the discomfort it can cause.

Mannitol has been shown to stimulate AVP release, but no study has tested copeptin levels after mannitol stimulation in healthy adults or patients with AVP-D or PP.

This single-center study is conducted in two consecutive parts. Part 1 is a double-blind, randomized cross-over proof-of-concept study in healthy adults to investigate if mannitol infusion stimulates copeptin release. Part 2 is an open-label, single arm case-control pilot study in adults with diagnosed PP or AVP-D to see if copeptin levels after mannitol stimulation differ in PP and AVP-D.

The results of this study aim to demonstrate if mannitol infusion has the potential to be used as an alternative to hypertonic saline infusion.

ELIGIBILITY:
Inclusion Criteria:

Part 1: Proof of Concept in Healthy adults

* Age ≥ 18 years
* Healthy with no medication except hormonal contraception

Part 2: Pilot Study in Patients with primary polydipsia (PP) or arginine vasopressin deficiency (AVP-D)

* Age ≥ 18 years
* Evidence of polyuria > 40-50 ml/kg body weight per 24 hours and polydipsia > 3 Liter per 24 hours or regular desmopressin medication corresponding to a diagnosis of PP or AVP-D

Exclusion Criteria:

Part 1: Proof of Concept in Healthy adults

* Participation in a trial with investigational drugs within 30 days
* Evidence of disordered drinking habits and diuresis defined as polyuria > 40-50 ml/kg body weight per 24 hours and polydipsia > 3 Liter per 24 hours.
* Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1,73 m2
* Glucose > 11.1 mmol/L corresponding to the diagnosis of an uncontrolled diabetes mellitus
* History of urinary tract obstruction
* Problems with urination
* Pregnancy or breastfeeding
* Multiple allergies (≥ 3)
* Evidence of acute illness

Part 2: Pilot Study in Patients with PP or AVP-D

* Participation in a trial with investigational drugs within 30 days
* Pregnancy or breastfeeding
* Evidence of acute illness
* eGFR < 60 ml/min/1,73 m2
* Glucose > 11.1 mmol/L corresponding to the diagnosis of uncontrolled diabetes mellitus
* History of urinary tract obstruction
* Problems with urination
* Therapy with diuretics
* Multiple allergies (≥ 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Difference in copeptin levels | Part 1: At 90 min post infusion, Part 2: at 30 min post infusion
  The difference in copeptin levels at 90 minutes following a 30-minute infusion of mannitol, part 1: compared to placebo in healthy adults and part 2: between patients with (primary polydipsia) PP and arginine vasopressin deficiency (AVP-D)

SECONDARY OUTCOMES:
Change of copeptin levels | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  Changes in copeptin levels compared to baseline.
Maximum copeptin levels | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  The maximum copeptin level after infusion is determined.
Assessment of hormone level | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in hormone levels, an assessment of hormones (e.g. Adrenocorticotropic hormone, Growth hormone, Insulin-like growth factor 1) is performed.
Assessment of serum electrolytes | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in electrolytes, an assessment of electrolytes (e.g. sodium potassium, chloride) in the serum is performed.
Assessment of plasma osmolality | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in parameters associated with fluid balance/ kidney function, an assessment of plasma osmolality (mOsm/kg) is performed.
Assessment of urea | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in parameters associated with fluid balance/ kidney function, an assessment of ureal levels (mmol/L) is performed.
Assessment of uric acid | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in parameters associated with fluid balance/ kidney function, an assessment of uric acid levels (umol/L) is performed.
Assessment of creatinine | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in parameters associated with fluid balance/ kidney function, an assessment of creatinine levels (umol/L) is performed.
Assessment of glucose | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change in parameters associated with fluid balance/ kidney function, an assessment of glucose levels (mmol/L) is performed.
Assessment of urine parameters | Part 1: At baseline, 90 and 150 min after infusion, Part 2: At baseline, 30 and 90 min after infusion
  To determine the change in urine parameters, an assessment of parameters (e.g. sodium, osmolality, creatinine) in the urine is performed.
Assessment of blood pressure | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change of vital parameters, the blood pressure (systolic and diastolic) is assessed.
Assessment of heart rate | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  To determine the change of vital parameters, the heart rate is assessed.
Assessment of adverse effects | Part 1: At baseline, 30, 45, 60, 90, and 150 min after infusion, Part 2: At baseline, 30 and 90 minutes
  The incidence of adverse effects, such as nausea, headache, fatigue, dizziness, thirst, is assessed using the numeric rating scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst possible pain."
Diagnostic accuracy of copeptin after mannitol Infusion for differentiating AVP-D from PP | Part 2: At 30 min post infusion
  Assessment of the diagnostic accuracy of stimulated copeptin levels measured after mannitol infusion to distinguish patients AVP-D from those with PP. The outcome will compare post-infusion copeptin concentrations between the two groups.
Assessment of changes in ECG QTc Interval | Part 2: at Baseline and 90 min after infusion
  Assessment of the change in the corrected QT (QTc) interval on a standard ECG
Assessment of changes in ECG Heart rate | Part 2: at Baseline and 90 min after infusion
  Assessment of the change in Heart rate on a standard ECG
Assessment of changes in ECG Cardiac rhythm | Part 2: at Baseline and 90 min after infusion
  Assessment of the change in Cardiac rhythm on a standard ECG
Assessment of changes in ECG QRS morphology | Part 2: at Baseline and 90 min after infusion
  Assessment of the change in QRS morphology on a standard ECG
Assessment of changes in ECG P- and T wave morphology | Part 2: at Baseline and 90 min after infusion
  Assessment of the change in P- and T wave morphology on a standard ECG

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland